CLINICAL TRIAL: NCT06832553
Title: The Effect of Surgical Incision Drep Use in Endotracheal Tube Fixation in Neonatal Preterm Infants: A Randomized Controlled Trial
Brief Title: The Effect of Surgical Incision Drep Use in Endotracheal Tube Fixation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Barış Çelik, Phd student, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024/101
Record Dates: First submitted 2024-12-07; First posted 2025-02-18 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Preterm
Keywords: preterm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Incision Drape (Experimental): Participants in this group will have their endotracheal tube (ETT) secured using a surgical incision drape. This method will be evaluated for its efficacy in preventing unplanned extubation and wound complications compared to the use of silk plasters.
  Interventions: Other: surgical incision drep
- silk plasters (Active Comparator): The endotracheal tube (ETT) of the participants in this group will be secured using silk plasters. This method will be evaluated for its efficacy in preventing unplanned extubation and wound complications compared to the use of a surgical incision drape.
  Interventions: Other: surgical incision drep

INTERVENTIONS:
Other: surgical incision drep — To compare the efficacy of surgical incision with silk plaster in ETT fixation.
  Other Names: silk plasters

SUMMARY:
It is aimed to minimise both unplanned extubation and skin damage with the surgical incision drep that we will use to fix the endotracheal tube in neonatal preterm infants and to reduce the complications that may develop due to these events. In addition, it is aimed to evaluate the relationship between these parameters by using devices measuring skin moisture, skin pH and Neonatal Skin Condition Assessment Scale in experimental and control groups.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effectiveness of surgical incision drape usage for securing endotracheal tubes in preterm neonates. The study will be conducted using a randomized controlled design, and participants will be divided into two groups: those using the surgical drape and those not using it. The population of the study will consist of preterm infants who are hospitalised in the neonatal intensive care unit of Batman Training and Research Hospital. Intubated preterm infants between 28-34 weeks will be included in the study regardless of gender difference. Research data will be collected by the following methods: Demographic information, Neonatal Skin Condition Rating Scale (NSCS), Skin Ph meter device and skin moisture meter device. Data will be collected every 24 hours during the intubation period. The results of the study are expected to provide important theoretical and practical contributions. The effects of parameters such as skin wounds that may occur due to endotracheal tube fixation in infants, unplanned extubation rates, skin pH and skin moisture at the site of intubation fixation will be compared between the surgical incision drep and the standard group. The research data will be analysed using IBM SPSS 27.0 Programme (Statistical Package for Social Sciences).

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants between 28-34 weeks of gestation hospitalized in neonatal intensive care unit,
* Intubated infants on invasive mechanical ventilators,
* Babies who were orally intubated were included in the study.

Exclusion Criteria:

* Congenital skin condition,
* With circulatory problems,
* Congenital anomalies and metabolic disorders,
* Small for gestational age (SGA) and large for gestational age (LGA),
* Unplanned extubation taking place,
* Babies intubated for less than 24 hours will be excluded from the study.

Ages: 28 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
demographic data | through study completion, an average of 1 year
  It will consist of questions such as gestational week, birth weight, postnatal age, frequency of endotracheal tube re-fixation, reason for hospitalization, frequency of aspiration, mode of delivery, gender, phototherapy status, antibiotic status, sedative use, analgesic use, ventilator mode.

SECONDARY OUTCOMES:
skin ph meter and skin moisture meter | through study completion, an average of 1 year
  During the intubation period, skin pH and skin moisture meter data will be obtained from the experimental and control group patients every 24 hours at the intubation fixation site.

OTHER OUTCOMES:
Newborn Skin Condition Assessment Scale | through study completion, an average of 1 year
  Data will be collected every 24 hours.The scale consists of three dimensions including dryness, redness and impaired skin integrity/peeling. The NSCS can be used in all newborns and a score between 3 and 9 is obtained. The lowest score of 3 indicates the best skin score, while the highest score of 9 indicates the worst skin score. skin wounds scores at the site of intubation tube fixation will be compared in experimental and control groups.
unplanned extubation | through study completion, an average of 1 year
  Data will be collected and statistical values will be calculated when an unplanned extubation event occurs in the experimental and control group patients while the patient is intubated.

CONTACTS AND LOCATIONS:
Overall Officials: Barış Çelik, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Barış Çelik, Batman, Turkey (Türkiye)